CLINICAL TRIAL: NCT03940807
Title: Phase III Trial to Assess Impact of Ultra-long Versus Long Down-regulation Protocol on IVF/ICSI Outcomes in Infertile Women Presenting With Adenomyosis.
Brief Title: Impact of Ultra-long Versus Long Down-regulation Protocol on IVF/ICSI in Adenomyosis
Acronym: ADENOFIV
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Principal investigator departure
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/17/0448
Record Dates: First submitted 2019-04-19; First posted 2019-05-07 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Adenomyosis
Keywords: Infertility; GnRH
MeSH Terms: conditions — Adenomyosis; Infertility | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra-long protocol group (Experimental): All women will receive one intra-muscular administration of 11.25 mg Gonadotropin Releasing Hormone (GnRH) agonist (triptorelin acetate) on luteal phase of their menstrual cycle. Add back therapy (transdermal estradiol, 25μg twice a week) will be administrated throughout down-regulation period. Ovarian stimulation will be started after 90 days desensitization.
  Interventions: Drug: 11.25mg GnRH agonist; Drug: 25 µg transdermal oestradiol
- Long protocol group (Active Comparator): All women will receive a 15-days pituitary down-regulation protocol that consists of daily subcutaneous application of 0.1mg of GnRH agonist (triptorelin acetate) started on luteal phase of their menstrual cycle. Ovarian stimulation will begin after 15 days desensitization.
  Interventions: Drug: 0.1 mg GnRH agonist

INTERVENTIONS:
Drug: 11.25mg GnRH agonist — Ultra-long protocol group women will receive one intra-muscular administration of 11.25 mg GnRH agonist (triptorelin acetate) on the luteal phase of their menstrual cycle. Ovarian stimulation will be started after 90 days desensitization.
  After the desensitization period, all patients will undergo standardized ovarian stimulation, follicular aspiration, fertilization of all oocytes using either standard insemination or ICSI according to the features of sperm examination, fresh embryo transfer and luteal phase support.
  Arms: Ultra-long protocol group
Drug: 0.1 mg GnRH agonist — Long protocol group women will receive a 15-days pituitary down-regulation protocol that consists of daily subcutaneous injection of 0.1mg of GnRH agonist (triptorelin acetate) started on the luteal phase of their menstrual cycle.
  Ovarian stimulation will begin after 15 days desensitization. After the desensitization period, all patients will undergo standardized ovarian stimulation, follicular aspiration, fertilization of all oocytes using either standard insemination or ICSI according to the features of sperm examination, fresh embryo transfer and luteal phase support.
  Arms: Long protocol group
Drug: 25 µg transdermal oestradiol — Add back therapy (transdermal estradiol, 25μg twice a week) will be administrated throughout down-regulation period.
  Arms: Ultra-long protocol group

SUMMARY:
Adenomyosis is a benign condition defined as the invasion of ectopic endometrium into the myometrium, resulting in smooth muscle hyperplasia and endometrial inflammation, commonly associated with endometriosis and uterine fibroids.

Heterogeneity among studies regarding diagnostic criteria and therapeutic management has fed the debate surrounding the impact of adenomyosis on assisted reproductive therapy outcomes. Nevertheless, recent data support that adenomyosis impairs reproductive outcomes associated with in vitro fertilization (IVF). According to several experimental data, prolonged exposure to gonadotropin releasing hormone (GnRH) agonists may overcome part of the detrimental impact of adenomyosis on fertility outcome. Overall, GnRH agonist treatment resulted in decreased local production of cytochrome P450 aromatase, decreased intrauterine concentration of free radicals and reduced inflammatory response and angiogenesis in endometrium, myometrium and adenomyosis lesions. At the same time, GnRH agonists affect neither endometrial capacity to support invasion nor invasive potential of the blastocyst in the early stages of implantation.

For IVF, 2 main protocols based on GnRH agonist pituitary down-regulation are available:

* the long protocol involving a 15 days pituitary down-regulation;
* the ultra-long protocol involving a 3 months pituitary down-regulation. Most studies using ultra-long protocol reported similar IVF outcomes in adenomyosis patients and control groups. Conversely, studies involving long or GnRH antagonist protocols demonstrated a significant reduction in clinical and ongoing pregnancy rates in adenomyosis patients compared to control subjects. Thus supporting that ultra-long protocol may be beneficial to improve IVF outcomes in the setting of adenomyosis.This is what investigators would like to demonstrate in this study

ELIGIBILITY:
Inclusion Criteria:

1. suspected adenomyosis on high quality transvaginal ultrasound or focal or diffuse adenomyosis defined as a thickening of the junctional zone to more than 12mm on previous magnetic resonance Imaging (<6 months)
2. infertility of any cause requiring IVF or ICSI
3. infertility period of at least 1 year except for women with history of deep infiltrating endometriosis or bilateral salpingectomy
4. age >18 and < 40 years
5. complete fertility workup comprising for women hormone serum measurement (anti-mullerian hormone (AMH), estradiol, follicle stimulating hormone (FSH), luteinizing hormone (LH)), high quality transvaginal ultrasound and, when applicable, hysterosalpingography, diagnostic laparoscopy or hysteroscopy
6. first or second IVF or ICSI attempt
7. absence of severe premature ovarian insufficiency defined by antral follicle count < 8 and AMH < 1ng/ml
8. meet the criteria from the French law to be included in an assisted reproductive technique program
9. informed written consent for both women and men
10. social security cover for both women and men

Exclusion Criteria:

1. absence of adenomyosis (defined as a thickening of the junctional zone to more than 12mm) on pelvic MRI
2. other potential causes of implantation failure: leiomyoma, endometrial polyp, not removed hydrosalpinx, malformed uterus (unicornis, bicornis, septate, duplex), antiphospholipid syndrome
3. medical contraindication to study treatments (GnRH agonist and add-back therapy)
4. women taking prohibited concomitant treatments and not able to stop them for the study period
5. medical contraindication to assisted reproductive technique and/or pregnancy including: uncontrolled type I and II diabetes; undiagnosed liver disease or dysfunction; renal insufficiency; history of deep venous thrombosis, pulmonary embolism or cerebrovascular accident; uncontrolled hypertension; known symptomatic heart disease; history of or suspected cervical carcinoma, endometrial carcinoma, ovarian carcinoma or breast carcinoma; undiagnosed vaginal bleeding; genetic abnormalities
6. positive plasma viral load for human immunodeficiency virus(HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV) for one (or both) in the couple during the year before inclusion
7. participation in another research study including an exclusion period which has not expired at the time of screening
8. patients subject to a judicial safeguard order, guardianship or trusteeship.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Number of live birth after first or second in vitro fertilization (IVF)/intra cytoplasmic sperm injection (ICSI) attempt. | Up to 22 weeks of gestation
  This outcome is defined as delivery of one or more live-born infant at > 22 weeks of gestation.

SECONDARY OUTCOMES:
Uterine volume change | after 90 days desensitization in ultra-long protocol group and after 15 days desensitization in long protocol group
  Uterine volume reduction between ultrasound measurements at baseline and at time of ovarian stimulation onset
Occurrence of poor responders | after 90 days desensitization in ultra-long protocol group and after 15 days desensitization in long protocol group
  Occurrence of poor responders defined as women with <3 matures follicles or serum estradiol <500 at the time of ovulation triggering
Concentration of serum Human Chorionic Gonadotropin (HCG or ßhCG) ≥ 100 IU/l | 14 days following follicular aspiration
  Biochemical pregnancy defined as serum Human Chorionic Gonadotropin (HCG or ßhCG) ≥ 100 IU/l, 14 days following follicular aspiration
Implantation rate | 5 weeks after follicular aspiration
  Implantation rate defined as the ratio "number of gestational sacs/number of transferred embryos" on TV US performed 5 weeks after follicular aspiration
Number of Participants with clinical pregnancy | 5 weeks after follicular aspiration
  Clinical pregnancy defined as the presence of one or more gestational sacs on transvaginal ultrasound performed 5 weeks after follicular aspiration, including ectopic pregnancy
Number of Participants with clinical pregnancy with fetal heart beat | 7 weeks after embryo transfer
  Clinical pregnancy with fetal heart beat defined as the presence of at least one fetus with heart beat on transvaginal ultrasound performed 7 weeks after embryo transfer
Number of Participants with ongoing pregnancy | 12 weeks of gestation
  Ongoing pregnancy defined as a live pregnancy on first trimester US examination performed at 12 weeks of gestation
First trimester miscarriage occurrence | Before 12 weeks of gestation
  First trimester miscarriage occurrence defined as a pregnancy loss before 12 weeks of gestation among patients with a clinical pregnancy
Occurrence of menopause-like symptoms symptoms at the end of the GnRH agonist treatment | after 90 days desensitization in ultra-long protocol group and after 15 days desensitization in long protocol group
  Using the Menopause Rating Scale
Occurrence of neonatal complications | Until 6 weeks post-partum
Occurrence of any other Adverse Event | Through study completion, an average of 1 year
Occurrence of pregnancy and post-partum complications | Until 6 weeks post-partum

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Vidal, Principal Investigator — University Hospital, Toulouse
Locations (14):
- France (14):
  - CHU Angers, Angers
  - Centre Aliénor d'Aquitaine, Bordeaux
  - Hôpital Morvan, Brest
  - Centre hospitalier intercommunal de Créteil, Créteil
  - CHU Grenoble-Alpes, Grenoble
  - CHU Limoges, Limoges
  - Hôpital de la Conception Marseille, Marseille
  - CHU Nice, Nice
  - CHU Nîmes, Nîmes
  - CHI Poissy, Poissy
  - CHU Rouen Normandie, Rouen
  - Centre hospitalier des 4 villes, Saint-Cloud
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No